CLINICAL TRIAL: NCT05830981
Title: Valproic Acid Use Evaluation in Patients With Neurological Disorders: a Retrospective and Prospective Analysis
Brief Title: Valproic Acid Use in Patients With Neurological Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damanhour University (Other)
Collaborators: Mansoura University (Other)
Responsible Party: Principal Investigator, Rehab Werida, Principal Investigator, Damanhour University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: valproic acid therapy
Record Dates: First submitted 2023-04-14; First posted 2023-04-26 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Neurological Disorders
Keywords: Valproate use
MeSH Terms: conditions — Nervous System Diseases | interventions — Early Intervention, Educational

STUDY DESIGN:
Intervention Model Description: A quasi-experimental pretest-posttest design study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phase 1 (No Intervention): n=600
- Phase 2 (Active Comparator): n=504
  Interventions: Other: Educational intervention

INTERVENTIONS:
Other: Educational intervention — 3 months of educational intervention (Lectures, information bulletin, handbook and hardcopy presentation slides) among professionals and patients.
  Other Names: Educational &counselling sessions
  Arms: Phase 2

SUMMARY:
Sodium valproate is a well-known anticonvulsant used in the treatment of epilepsy and bipolar disorder, as well as other psychiatric conditions requiring the administration of mood stabilizers. Aim of the present study is to assess sodium valproate usage among patients with neurological disorders.

Prescriptions of 600 patients from out-patient pharmacy of neurology department at Mansoura university teaching hospital were analyzed in a retrospective prospective observational study which conducted between January 2015 and December 2017. Data collected include: demographic data, medical history, drug-drug interaction, polypharmacy, medication error, doses and therapeutic duplication. A designed and structured form was used to collect the required information.

DETAILED DESCRIPTION:
This quasi-experimental pretest-posttest design study was conducted at the outpatient's pharmacy of Neurology department at tertiary care hospital. After identifying problems with use and completing a follow-up, 3 months of educational intervention (Lectures) among professionals was given. As this study is observational informed consent from all subjects was waived. The subjects were enrolled on the basis of inclusion and exclusion criteria. Patients receiving at least 7 days of Valproic acid, between 10-70 years old, both sexes, were included in the study figure 1. 600 Prescriptions were reviewed between January of 2015 to December of 2017 for patients who were suffering from any psychotic illness and were on psychiatric medications. Then pharmacist educational intervention started and followed up for three months then prescriptions re-evaluted.

Inclusion/ exclusion criteria: The study population was limited to those who were continuously eligible for the outpatient pharmacy refilling thier medications during the entire study period. Patients were identified through pharmacy drug prescriptions By hospital policy all drugs are prescribed for a maximum period of 3 months. Consequently, all patients presented at least twice during the study period. A designed and structured form was used to collect the required information. Data then collected on Microsoft Excel sheet, which included patients' initial therapeutic indications, concomitant use of oral medications, significant adverse drug effects and any drug -drug interaction.

ELIGIBILITY:
Inclusion Criteria:

* The study population was limited to those who prescribed with valproate and were continuously eligible for the outpatient during the entire study period. Patients were identified through pharmacy drug prescriptions By hospital policy all drugs are prescribed for a maximum period of 3 months. Consequently, all patients presented at least twice during the study period.

Exclusion Criteria:

* Patients who not use valproate.

Ages: 10 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2017-12-20 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Valproate dose (Number) | 3 month
  Right dose
Number of drugs (Number) | 3 Months
  Number of drugs included in the prescriptions analyzed
Medication errors (Number) | 3 Months
  Medication errors regarding frequency or dose of Sodium valproate
Adherence (Number) | 3 Months
  Adherence to medication regimens
Tolerability (Number) | 3 Months
  tolerability was assessed through monitoring of ADRs and recorded in the patient's file.

CONTACTS AND LOCATIONS:
Overall Officials: Rehab H Werida, Ass. Prof., Principal Investigator — Damanhour University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thakkar KB, Jain MM, Billa G, Joshi A, Khobragade AA. A drug utilization study of psychotropic drugs prescribed in the psychiatry outpatient department of a tertiary care hospital. J Clin Diagn Res. 2013 Dec;7(12):2759-64. doi: 10.7860/JCDR/2013/6760.3885. Epub 2013 Dec 15. PMID 24551631
- [Background] Bell JS, Whitehead P, Aslani P, McLachlan AJ, Chen TF. Drug-related problems in the community setting: pharmacists' findings and recommendations for people with mental illnesses. Clin Drug Investig. 2006;26(7):415-25. doi: 10.2165/00044011-200626070-00003. PMID 17163274
- [Background] Nanaumi Y, Yoshitani A, Onda M. Impact of interventions by a community pharmacist on care burden for people with dementia: development and randomized feasibility trial of an intervention protocol. Pilot Feasibility Stud. 2022 Jun 2;8(1):118. doi: 10.1186/s40814-022-01071-7. PMID 35655244
- [Derived] Werida RH, El-Sherif S, Shoshan R, Khedr NF. Evaluation of prescribing patterns of sodium valproate in neurological disease patients: a quasi-experimental pretest-posttest design study. BMC Health Serv Res. 2025 Mar 27;25(1):441. doi: 10.1186/s12913-025-12483-5. PMID 40140829